CLINICAL TRIAL: NCT00844298
Title: Tasigna® (Nilotinib) Plus Multi-Agent Chemotherapy for Newly-Diagnosed Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia
Brief Title: Nilotinib and Combination Chemotherapy in Treating Patients With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Kyoo-Hyung Lee, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000632225; AMC-UUCM-2008-0310; NOVARTIS-AMC-UUCM-2008-0310
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Leukemia
Keywords: Philadelphia chromosome positive adult precursor acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Rituximab; Asparaginase; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nilotinib+mVPD (Experimental): Patients who were Philadelphia-positive, newly-diagnosed adult ALL and treated with nilotinib + mVPD treatment plan
  Interventions: Drug: Nilotinib+mVPD

INTERVENTIONS:
Drug: Nilotinib+mVPD — 1. Induction:
     * Daunorubicin 90 mg/m2/day by continuous iv infusion (d1-3)
     * Vincristine 2 mg iv push (d1, 8, 15, 22)
     * Prednisolone 60 mg/m2/day po (d1-28)
     * Nilotinib 400mg bid/d (d8-)
  2. Consolidation A (cycle1)
     * Daunorubicin 45 mg/m2/day by continuous iv (d1, 2)
     * Vincristine 2 mg iv (d1, 8)
     * Prednisolone 60 mg/m2/day po (d1-14)
     * Nilotinib 400mg bid/d
  3. Consolidation B (cycles 2&4)
     * Cytarabine 2,000 mg/m2/day iv over 2 hours (d1-4)
     * Etoposide 150 mg/m2/day iv over 3 hours (d1-4)
     * Nilotinib 400mg bid/d
  4. Consolidation C (cycles 3&5)
     * Methotrexate 220 mg/m2 iv bolus, then 60mg/m2/h for 36 hours (d1-2, 15-16)
     * Leucovorin followed immediately by 50 mg/m2 iv every 6hrs for three doses,
     * Nilotinib 400mg bid/d
  5. Maintenance
     ◦Nilotinib 400mg bid/d (during 2 years, for patients without alloHCT)
  6. Consider alloHCT
  Other Names: Mabthera; VCS; Daunobrastina; Solondo; Leunase; Cytarabine; Efosin; DBLMethotrexate

SUMMARY:
RATIONALE: Nilotinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving nilotinib together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving nilotinib together with combination chemotherapy works in treating patients with newly diagnosed acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the clinical efficacy of nilotinib and combination chemotherapy, in terms of hematologic and molecular complete remission (CR) rates, in patients with newly diagnosed Philadelphia chromosome-positive acute lymphoblastic leukemia or acute mixed lineage leukemia.

Secondary

* To establish the prognostic factors for patients treated with this regimen.
* To determine the duration of CR in patients treated with this regimen.
* To determine the duration of progression-free and overall survival of these patients.
* To determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to age (15 to 64 years vs ≥ 65 years).

* Induction therapy: Patients receive daunorubicin hydrochloride IV continuously over 24 hours on days 1-3, vincristine sulfate IV on days 1 and 8, and oral prednisolone on days 1-14. Patients undergo bone marrow examination on day 14. Patients in hematologic remission proceed to consolidation therapy. Patients with residual leukemic cells > 5% receive an additional dose of daunorubicin hydrochloride IV continuously over 24 hours on day 15 before proceeding to consolidation therapy.
* Consolidation therapy: For course 1, patients receive daunorubicin hydrochloride IV continuously over 24 hours on days 1 and 2, vincristine sulfate IV on days 1 and 8, and oral prednisolone on days 1-14. For courses 2 and 4, patients receive cytarabine IV over 2 hours and etoposide IV over 3 hours on days 1-4. For courses 3 and 5, patients receive methotrexate IV continuously over 36 hours on days 1, 2, 15, and 16 and leucovorin calcium IV every 6 hours for 3 doses and then orally until blood methotrexate levels are in a safe range.

Patients also receive oral nilotinib twice daily beginning on day 8 of induction therapy and continuing until the completion of consolidation therapy.

After completion of consolidation therapy, patients with a hematopoietic stem cell donor proceed to allogeneic hematopoietic stem cell transplantation (HSCT). Patients who do not undergo HSCT continue to receive oral nilotinib twice daily for up to 2 years after completion of consolidation therapy.

After completion of study therapy, patients are followed periodically for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute lymphoblastic leukemia or acute mixed lineage leukemia

  * Positive for Bcr-Abl fusion transcript (Philadelphia chromosome-positive disease) by RT-PCR

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Total bilirubin < 2 mg/dL
* SGOT < 3 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN (unless considered tumor-related)
* Creatinine < 2.0 mg/dL ULN
* Serum amylase and lipase ≤ 1.5 times ULN
* Potassium, magnesium, and phosphorus normal (supplementation allowed)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No rare hereditary problems with galactose intolerance, severe lactase deficiency, or glucose-galactose malabsorption
* No known sensitivity to any of the study drugs
* No severe medical condition that, in the opinion of the investigator, would preclude study participation
* No impaired cardiac function, including any of the following:

  * LVEF < 45% or below the lower limit of normal by ECHO
  * Long QT syndrome or known family history of long QT syndrome
  * Clinically significant resting bradycardia (< 50 beats per minute)
  * QTc > 450 msec on baseline ECG (using the QTcF formula)
  * Myocardial infarction within the past 12 months
  * Other clinically significant heart disease, including any of the following:

    * Unstable angina
    * Congestive heart failure
    * Uncontrolled hypertension
    * Uncontrolled arrhythmias
* No other primary malignant disease requiring systemic treatment
* No acute or chronic liver, pancreatic, or severe renal disease
* No other severe and/or life-threatening medical disease
* No history of significant congenital or acquired bleeding disorder unrelated to cancer
* No impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug
* No history of non-compliance

PRIOR CONCURRENT THERAPY:

* More than 30 days since prior investigational agents
* No concurrent medications that have the potential to prolong the QTc interval
* No concurrent strong CYP3A4 inhibitors
* No concurrent therapeutic coumarin derivatives

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-01; Primary Completion 2012-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoo H. Lee, MD, Principal Investigator — Asan Medical Center
Locations (16):
- South Korea (16):
  - Daegu Fatima Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Daegu Catholic University Hospital, Daegu
  - National Cancer Center - Korea, Goyang
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Gyeongsang National University Hospital, Jinju
  - Pusan National University Hospital, Pusan
  - Inje University Seoul Paik Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center - University of Ulsan College of Medicine, Seoul
  - Konkuk University Medical Center, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Kim DY, Joo YD, Lim SN, Kim SD, Lee JH, Lee JH, Kim DH, Kim K, Jung CW, Kim I, Yoon SS, Park S, Ahn JS, Yang DH, Lee JJ, Lee HS, Kim YS, Mun YC, Kim H, Park JH, Moon JH, Sohn SK, Lee SM, Lee WS, Kim KH, Won JH, Hyun MS, Park J, Lee JH, Shin HJ, Chung JS, Lee H, Eom HS, Lee GW, Cho YU, Jang S, Park CJ, Chi HS, Lee KH; Adult Acute Lymphoblastic Leukemia Working Party of the Korean Society of Hematology. Nilotinib combined with multiagent chemotherapy for newly diagnosed Philadelphia-positive acute lymphoblastic leukemia. Blood. 2015 Aug 6;126(6):746-56. doi: 10.1182/blood-2015-03-636548. Epub 2015 Jun 11. PMID 26065651

RESULTS

PARTICIPANT FLOW:
Groups:
- Nilotinib+mVPD: Patients who were Philadelphia-positive, newly-diagnosed adult ALL and treated with nilotinib + mVPD treatment plan
  Nilotinib+mVPD: 1.Induction:
  * Daunorubicin 90 mg/m2/day by continuous iv infusion (d1-3)
  * Vincristine 2 mg iv push (d1, 8, 15, 22)
  * Prednisolone 60 mg/m2/day po (d1-28)
  * Nilotinib 400mg bid/d (d8-) 2.Consolidation A (cycle1)
  * Daunorubicin 45 mg/m2/day by continuous iv (d1, 2)
  * Vincristine 2 mg iv (d1, 8)
  * Prednisolone 60 mg/m2/day po (d1-14)
  * Nilotinib 400mg bid/d
    3. Consolidation B (cycles 2&4)
  * Cytarabine 2,000 mg/m2/day iv over 2 hours (d1-4)
  * Etoposide 150 mg/m2/day iv over 3 hours (d1-4)
  * Nilotinib 400mg bid/d
    4.Consolidation C (cycles 3&5)
  * Methotrexate 220 mg/m2 iv bolus, then 60mg/m2/h for 36 hours (d1-2, 15-16)
  * Leucovorin followed immediately by 50 mg/m2 iv every 6hrs for three doses,
  * Nilotinib 400mg bid/d
    5.Maintenance
  * Nilotinib 400mg bid/d (during 2 years, for patients without alloHCT)
    6.Consider alloHCT
Period: Overall Study
Arm/Group | Nilotinib+mVPD
Started | 91
Completed | 91
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nilotinib+mVPD
Number analyzed (Participants) | 90
Age, Continuous [Median (Full Range); unit: years] | 47.0 [17 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 45

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving Hematologic and Molecular Complete Remission (CR) After Induction Therapy
Description: approximate time: at the recovery of cytopenia
Time Frame: 1 month
Measure: Number; unit: percentage of analyzable subjects
Arm/Group | Nilotinib+mVPD
Number analyzed (Participants) | 90
percentage of analyzable subjects | 91

2. Secondary Outcome: Disease(Relapse)-Free Survival
Time Frame: 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Nilotinib+mVPD
Serious Adverse Events (participants affected / at risk) | 18/91
Other Adverse Events (participants affected / at risk) | 79/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib+mVPD (N=91)
Febrile neutropenia (Infections and infestations) | 18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nilotinib+mVPD (N=91)
Jaundice (Hepatobiliary disorders) | 79 (214)

LIMITATIONS AND CAVEATS:
The limitation of the current study was that this study was not performed in a randomized comparative way, and the advantages of nilotinib over other TKIs were not definitely demonstrated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No